CLINICAL TRIAL: NCT00331409
Title: A Phase II Study of the Mammalian Target of Rapamycin (mTOR) Inhibitor RAD001 in Combination With Imatinib Mesylate in Patients With Previously Treated Advanced Renal Carcinoma
Brief Title: Everolimus and Imatinib Mesylate in Treating Patients With Metastatic or Unresectable Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christopher Ryan, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00001754; OHSU-SOL-05108-LM (Other: OHSU Knight Cancer Institute); FWA00000161 (Other: OHSU IRB); OHSU-1754 (Other: OHSU IRB); CDR0000479150 (Other: NCI PDQ)
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Results first posted 2011-10-05 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-09

CONDITIONS: Kidney Cancer
Keywords: stage III renal cell cancer; stage IV renal cell cancer; clear cell renal cell carcinoma; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Everolimus; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus and Imatinib Mesylate (Experimental): Everolimus: 2.5 mg daily by mouth Imatinib Mesylate: 600 mg daily by mouth
  Interventions: Drug: Everolimus; Drug: imatinib mesylate

INTERVENTIONS:
Drug: Everolimus — 2.5 mg by mouth daily
  Other Names: Afinitor; RAD001; Certican
Drug: imatinib mesylate — 600 mg by mouth daily
  Other Names: Gleevec; STI-571

SUMMARY:
RATIONALE: Everolimus and imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Everolimus may also block blood flow to the tumor. Giving everolimus together with imatinib mesylate may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving everolimus together with imatinib mesylate works in treating patients with metastatic or unresectable kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the proportion of patients with previously treated metastatic or unresectable clear cell carcinoma of the kidney who are progression free (complete response [CR], partial response [PR], or stable disease [SD]) at 3 months after treatment with everolimus and imatinib mesylate.

Secondary

* Estimate median time to progression in patients treated with this regimen.
* Determine the proportion of patients whose best overall response are CR, PR, SD, or progressive disease.
* Evaluate the mean and range of the maximum percent reduction in tumor size.
* Describe the toxicities of this regimen in these patients.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral imatinib mesylate and oral everolimus once daily beginning on day 1 and continuing in the absence of disease progression.

PROJECTED ACCRUAL: A total of 43 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed clear cell kidney cancer, meeting 1 of the following criteria:

  * Measurable metastatic disease
  * Locally unresectable disease
* No history of known brain metastases that have not been adequately treated with radiotherapy and/or surgery
* Must have received ≥ 1 prior systemic therapy for metastatic or unresectable renal cell carcinoma

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 8 g/dL
* Bilirubin < 1.5 times upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase(SGOT) and Serum glutamic pyruvic transaminase(SGPT) < 2.5 times ULN
* Creatinine < 1.5 times ULN
* No New York Heat Association grade III-IV cardiac disease
* No other malignancy within the past 5 years except basal cell skin cancer, cervical carcinoma in situ, or insignificant or inactive disease
* No chronic liver disease (i.e., chronic active hepatitis or cirrhosis)
* No severe or uncontrolled medical disease
* No gastrointestinal disease or impairment that would hinder the absorption of everolimus
* No uncontrolled diabetes
* No chronic renal disease
* No active uncontrolled infection
* No congestive heart failure
* No myocardial infarction within the past 6 months

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 2 weeks since prior major surgery
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosourea or mitomycin C)
* More than 4 weeks since prior immunotherapy
* More than 4 weeks since other prior investigational agents
* No prior radiotherapy to > 25% of bone marrow
* No prior treatment with an mammalian target of rapamycin(mTOR) inhibitor
* No concurrent therapeutic warfarin

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W. Ryan, MD, Study Chair — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initial recruitment began in Feb 2006 and ended in Dec 2007. 19 patients were put on study during that time frame. These patients came from OHSU oncology clinics or referrals to OHSU.
Pre-assignment Details: During the first stage, patients not assessable for progression-free status at 3 months due to study discontinuation for any reason except death or progression were replaced only for purposes of determining continuation to the second stage.A total of 19 patients were enrolled in the first stage 15 evaluable patients and 4 patients who were not.
Period: Overall Study
Arm/Group | Everolimus and Imatinib Mesylate
Started | 19 (19 patients were enrolled in the first stage due to 4 patients who withdrew early.)
Completed | 15 (15 patients accrued to the first stage;if>9 were progression-free at 3 months,enrollment continued.)
Not Completed | 4
Not completed — Lack of Efficacy | 4

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus and Imatinib Mesylate
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (7.7459)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 19

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival at 3 Months
Time Frame: 3 months post 1st dose
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus and Imatinib Mesylate
Number analyzed (Participants) | 19
months | 2.9 [1.9 to 6.2]

2. Primary Outcome: Overall Number of Participants Who Achieve a Response Rate (Complete Response, Partial Response, and Stable Disease) at 3 Months
Time Frame: Up to 4 years
Measure: Number; unit: participants
Arm/Group | Everolimus and Imatinib Mesylate
Number analyzed (Participants) | 19
participants | 18

3. Secondary Outcome: Median Time to Progression
Time Frame: Time to progression
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Everolimus and Imatinib Mesylate
Number analyzed (Participants) | 19
months | 2.9 [1.9 to 6.2]

4. Secondary Outcome: Number of Subjects That Demonstrated a Reduction in Tumor Measurements.
Description: Number of subjects that received at least one post-baseline scan that demonstrated a reduction in sum target lesions per Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
Time Frame: Up to 4 years
Population: 2 subjects were not evaluable. Reduction in target lesion sum did not meet the criteria for Partial Response (PR) for any of the subjects. Partial Response, per RECIST, includes at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD.
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus and Imatinib Mesylate
Number analyzed (Participants) | 17
Participants | 5

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Toxicity assessments will be obtained as follows:
  Cycle 1: Weeks 1,2,3 Cycle 2: Weeks 6,9 Cycle 3: Weeks 12, 15 Cycle 4: Weeks 18, 21 Cycle 5: Weeks 24, 27 Cycle 6+: Every visit during these cycles
  Safety assessments will consist of evaluating adverse events and serious adverse events.
Time Frame: Duration of study, Up to 4 years
Measure: Number; unit: participants
Arm/Group | Everolimus and Imatinib Mesylate
Number analyzed (Participants) | 19
participants | 19

ADVERSE EVENTS:
Arm/Group | Everolimus and Imatinib Mesylate
Serious Adverse Events (participants affected / at risk) | 10/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus and Imatinib Mesylate (N=19)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1
Pleural Effusions (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis (Infections and infestations) | 1
Fatigue (General disorders) | 2
Angioedema Tongue (Blood and lymphatic system disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Syncope (Vascular disorders) | 1
Hypotension (Cardiac disorders) | 1
Renal Failure (Renal and urinary disorders) | 1
Urinary Tract Infrection (Infections and infestations) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Periorbital Edema (Blood and lymphatic system disorders) | 1 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus and Imatinib Mesylate (N=19)
Decreased Hematrocrit (Blood and lymphatic system disorders) | 1
Decreased Hemoglobin (Blood and lymphatic system disorders) | 6 (6)
Decreased Lymphocytes (Blood and lymphatic system disorders) | 1
Decreased Platelet Count (Blood and lymphatic system disorders) | 2 (2)
Increased Bun (Blood and lymphatic system disorders) | 1 (1)
Low Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
Low Platelet Count (Blood and lymphatic system disorders) | 3 (3)
Low White Blood Cell Count (Blood and lymphatic system disorders) | 2 (2)
Lymphomenia (Blood and lymphatic system disorders) | 1 (1)
Lymphopemia (Blood and lymphatic system disorders) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Bradycardia (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 2 (2)
Mild congestive heart failure (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Unstable angina (Cardiac disorders) | 1 (1)
Chills/Rigors (General disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Fever (General disorders) | 4 (4)
Insomnia (General disorders) | 1 (1)
Weight Loss (General disorders) | 3 (3)
Abrasions: face, chest, arm (Skin and subcutaneous tissue disorders) | 1 (1)
Allergic reaction: hives (Skin and subcutaneous tissue disorders) | 1 (1)
Bruising on Abdomen (Skin and subcutaneous tissue disorders) | 1 (1)
Diabetic ulcer: toe (Skin and subcutaneous tissue disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1)
FACIAL FLUSHING (Skin and subcutaneous tissue disorders) | 2 (2)
ANOREXIA (Metabolism and nutrition disorders) | 13 (13)
Dehydration (Gastrointestinal disorders) | 4
Dysgeusia (Gastrointestinal disorders) | 2
Dysguesia (Gastrointestinal disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 4
NAUSEA (Gastrointestinal disorders) | 15
Hematuria (Blood and lymphatic system disorders) | 3
Muscles weakness (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 1
Abdominal Pain (General disorders) | 3

LIMITATIONS AND CAVEATS:
Our phase II study closed after the first stage of accrual due to an insufficient number of participants who remained progression-free at 3 months, per the study design.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No